CLINICAL TRIAL: NCT02098005
Title: A Modern Neuroscience Approach to Chronic Spinal Pain: Pain Neuroscience Education Combined With Cognition-targeted Motor Control Training
Brief Title: Pain Neuroscience Education Combined With Cognition-targeted Motor Control Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other); Vrije Universiteit Brussel (Other); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC/2013/1133
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Chronic Spinal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): usual care evidence-based physiotherapy
  Interventions: Other: usual care evidence-based physiotherapy
- modern neuroscience approach (Experimental): modern neuroscience approach
  Interventions: Other: modern neuroscience approach

INTERVENTIONS:
Other: usual care evidence-based physiotherapy — Arm 1 (i.e., the control group) will be subjected to a control intervention, including back/neck school and general exercises. 3 sessions of education (session 1: group session; session 2: online module; session 3: individual session) will be given by a physiotherapist, followed by 15 sessions of traditional physiotherapy and general exercises. The 18 sessions will be spread over a period of 3 months.
  Arms: Usual care
Other: modern neuroscience approach — Arm 2 (i.e., the experimental group) will receive pain neuroscience education (3 sessions of education), followed by 15 sessions of cognition-targeted motor control training (15 sessions). The 18 sessions will be spread over a period of 3 months.
  Arms: modern neuroscience approach

SUMMARY:
Chronic spinal pain (CSP) includes chronic low back pain, failed back surgery, chronic whiplash associated disorders, chronic non-traumatic neck pain, etc. The current investigators and others have provided evidence for impaired motor control of spinal muscles in patients with CSP. In addition, there is increasing evidence that central mechanisms, i.e. hyperexcitability of the central nervous system and brain abnormalities (e.g. decreased brain matter density) play a role in CSP. Hence, treatments for CSP should not only address the spinal muscles and joints, but also the brain. Therefore, a modern neuroscience approach, comprising of pain neuroscience education followed by cognition-targeted motor control training, can be applied.

The scientific objective entails examining the effectiveness of the modern neuroscience approach vs. usual care evidence-based physiotherapy for reducing pain and improving functioning in Flemish patients with CSP. A secondary objective entails examining the effectiveness of the modern neuroscience approach vs. usual care evidence-based physiotherapy for altering brain's structure and function (magnetic Resonance Imaging) in Flemish patients with CSP. Therefore, a multi-center triple-blind randomized controlled trial will be conducted.

To comply with this scientific objective, 120 CSP patients will be recruited and subjected to the baseline assessment. The baseline assessment includes the assessment of pain (including symptoms of central sensitization and conditioned pain modulation), the assessment of restrictions in functioning, brain imaging, the evaluation of motor control and muscle properties, spinal mobility, and psychosocial correlates. Baseline analysis will provide descriptive statistics and will lead to calculate correlation between the different outcome measures and predictors of pain and dysfunctioning. In a next step, included patients will be randomized to the experimental or control group. Those in the experimental group will receive neuroscience education combined with cognition-targeted motor control training. Those in the control group will be subjected to a control intervention, including back/neck school and general exercises. After the neuroscience education has been given, the experimental subjects will fill in the neurophysiology of pain test. Several follow-up assessments will take place. Part of the assessment (functionality (PDI questionnaire) and psychosocial correlates (Pain Catastrophizing Scale (PCS), pain vigilance and awareness questionnaire (PVAQ), Tampa Scale for Kinesiophobia (TSK), Illness Perception Questionnaire revised (IPQ-R)) will be re-evaluated after the first 3 sessions. The complete 'baseline' assessment will be repeated in the month following the treatment complement, rounding up the short-term follow-up assessment. Six months after the baseline assessment, pain, functioning and psychological correlates are assessed in an intermediate online assessment. One year after baseline assessment the complete assessment is repeated for the last time, unless the intermediate assessment indicates that treatment effects are no longer present. Both short and long term treatment effects can be studied and predictors for therapy success can be unraveled. Also correlations between changes in different outcome measures can provide relevant and innovative information.

The proof of principal suggests a strong effect reported by large effect sizes for pain and disability compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific spinal pain of at least 3 months' duration, at least 3 days per week
* Aged between 18 and 65 years
* Seeking care because of neck pain or low back pain
* Living or working within a radius of 50 km around the therapy location
* Not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain a steady state)
* Nonspecific failed back surgery > 3 years are permitted
* Not undertaking exercise (> 3 metabolic Equivalents) 3 days before the experiment
* Refraining from analgesics 48h prior to assessments.
* Abstaining from caffeine, alcohol or nicotine 24h prior to assessment

Exclusion Criteria:

* Neuropathic pain
* Chronic widespread pain
* Being pregnant or having given birth in the preceding year
* Contra-indications related to MRI imaging
* History of specific spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment (questionnaire) | at baseline
  questionnaire: numerical rating scale (NRS), central sensitization inventory (CSI), medical outcomes short form 36 health service (SF-36)
Pain assessment (physical testing) | at baseline
  Physical testing: pressure pain threshold (PTT), cold pressor test (CPT)
Functional assessment (questionnaires) | at baseline
  Questionnaires: PDI, SF-36
Pain assessment (questionnaire) | at 3 months
  questionnaire: numerical rating scale (NRS), central sensitization inventory (CSI), medical outcomes short form 36 health service (SF-36) Time Frame: after 18 treatment sessions
Pain assessment (questionnaire) | at 6 months
  questionnaire: numerical rating scale (NRS), central sensitization inventory (CSI), medical outcomes short form 36 health service (SF-36)
Pain assessment (questionnaire) | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  questionnaire: numerical rating scale (NRS), central sensitization inventory (CSI), medical outcomes short form 36 health service (SF-36)
Pain assessment (physical testing) | at 3 months
  Physical testing: pressure pain threshold (PTT), cold pressor test (CPT) Time Frame: after 18 treatment sessions
Pain assessment (physical testing) | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  Physical testing: pressure pain threshold (PTT), cold pressor test (CPT)
Functional assessment (questionnaires) | at 1 week
  Questionnaires: PDI, SF-36 Timeframe: after 3 treatment sessions (PDI)
Functional assessment (questionnaires) | at 3 months
  Questionnaires: PDI, SF-36 Time Frame: after 18 treatment sessions
Functional assessment (questionnaires) | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  Questionnaires: PDI, SF-36
Functional assessment (questionnaires) | at 6 months
  Questionnaires: PDI, SF-36

SECONDARY OUTCOMES:
Gray and white matter structure | at baseline
  Gray and white matter structure and function in brain areas involved in pain processing and sensorimotor control.
  Gray matter density - gray matter volumes - cortical thickness - surface area. Integrity of the white matter circuitry (tractography) - structural white matter connectivity - fractional anisotropy Intrinsic brain activity (cortex and nuclei) - functional connectivity
Motor Control | at baseline
  1. Postural steadiness
  2. Habitual standing posture
  3. Spinal range of motion
  4. Sensorimotor control
  i. Proprioception: position-reposition accuracy ii. Neuromuscular control (patients' ability to perform the skill of activation of specific, deep stabilizing muscles iii. Movement control of the spine
Psychological correlates | at baseline
  Psychological correlates: PCS, PVAQ, TSK, IPQ-R
Neurophysiology of pain test (questionnaire) | at 1 week
  Time Frame: after 3 treatment sessions Questionnaire: Dutch Neurophysiology of Pain Test (patient version)
Psychological correlates | at 1 week
  Psychological correlates: PCS, PVAQ, TSK, IPQ-R Time Frame: after 3 treatment sessions
Psychological correlates | at 3 months
  Psychological correlates: PCS, PVAQ, TSK, IPQ-R Time Frame: after 18 treatment sessions
Psychological correlates | at 6 months
  Psychological correlates: PCS, PVAQ, TSK, IPQ-R
Psychological correlates | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  Psychological correlates: PCS, PVAQ, TSK, IPQ-R
Muscle properties | at baseline
  1. Isometric muscle strength of spinal flexor and extensor muscles
  2. Endurance of spinal flexor and extensor muscles
Muscle properties | at 3 months
  1. Isometric muscle strength of spinal flexor and extensor muscles
  2. Endurance of spinal flexor and extensor muscles
  Time Frame: after 18 treatment sessions
Muscle properties | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  1. Isometric muscle strength of spinal flexor and extensor muscles
  2. Endurance of spinal flexor and extensor muscles
Motor Control | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  1. Postural steadiness
  2. Habitual standing posture
  3. Spinal range of motion
  4. Sensorimotor control
  i. Proprioception: position-reposition accuracy ii. Neuromuscular control (patients' ability to perform the skill of activation of specific, deep stabilizing muscles iii. Movement control of the spine
Motor Control | at 3 months
  1. Postural steadiness
  2. Habitual standing posture
  3. Spinal range of motion
  4. Sensorimotor control
  i. Proprioception: position-reposition accuracy ii. Neuromuscular control (patients' ability to perform the skill of activation of specific, deep stabilizing muscles iii. Movement control of the spine
  Time Frame: after 18 treatment sessions
Gray and white matter structure | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  Gray and white matter structure and function in brain areas involved in pain processing and sensorimotor control.
  Gray matter density - gray matter volumes - cortical thickness - surface area. Integrity of the white matter circuitry (tractography) - structural white matter connectivity - fractional anisotropy Intrinsic brain activity (cortex and nuclei) - functional connectivity
Gray and white matter function | at 3 months
  Gray and white matter structure and function in brain areas involved in pain processing and sensorimotor control.
  Gray matter density - gray matter volumes - cortical thickness - surface area. Integrity of the white matter circuitry (tractography) - structural white matter connectivity - fractional anisotropy Intrinsic brain activity (cortex and nuclei) - functional connectivity
  Time Frame: after 18 treatment sessions
Gray and white matter structure | at 3 months
  Gray and white matter structure and function in brain areas involved in pain processing and sensorimotor control.
  Gray matter density - gray matter volumes - cortical thickness - surface area. Integrity of the white matter circuitry (tractography) - structural white matter connectivity - fractional anisotropy Intrinsic brain activity (cortex and nuclei) - functional connectivity
  Time Frame: after 18 treatment sessions
Gray and white matter function | at 12 months (except when no treatment effects would be found at 6 months: go/no go principle)
  Gray and white matter structure and function in brain areas involved in pain processing and sensorimotor control.
  Gray matter density - gray matter volumes - cortical thickness - surface area. Integrity of the white matter circuitry (tractography) - structural white matter connectivity - fractional anisotropy Intrinsic brain activity (cortex and nuclei) - functional connectivity
Gray and white matter function | at baseline
  Gray and white matter structure and function in brain areas involved in pain processing and sensorimotor control.
  Gray matter density - gray matter volumes - cortical thickness - surface area. Integrity of the white matter circuitry (tractography) - structural white matter connectivity - fractional anisotropy Intrinsic brain activity (cortex and nuclei) - functional connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Danneels, MD, PhD, Principal Investigator — University Ghent; Jo Nijs, MD, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (3):
- Belgium (3):
  - Ghent University Hospital, Ghent
  - Universiteit Gent (UGent), Faculty of Medicine and Health Sciences, Dpt. Of Rehabilitation Sciences and Physiotherapy, BE-9000 Gent (Belgium), Ghent
  - Vrije Universiteit Brussel, Faculty of Physical Education & Physiotherapy, Dpt. of Rehabilitation Sciences & Physiotherapy, Jette

REFERENCES:
- [Derived] Van Bogaert W, Liew BXW, Fernandez-de-Las-Penas C, Valera-Calero JA, Varol U, Coppieters I, Kregel J, Nijs J, Meeus M, Cagnie B, Danneels L, Malfliet A. Exploring Interactions Between Sex, Pain Characteristics, Disability, and Quality of Life in People With Chronic Spinal Pain: A Structural Equation Model. J Pain. 2024 Mar;25(3):791-804. doi: 10.1016/j.jpain.2023.10.010. Epub 2023 Oct 21. PMID 37871684
- [Derived] Van Bogaert W, Coppieters I, Kregel J, Nijs J, De Pauw R, Meeus M, Cagnie B, Danneels L, Malfliet A. Influence of Baseline Kinesiophobia Levels on Treatment Outcome in People With Chronic Spinal Pain. Phys Ther. 2021 Jun 1;101(6):pzab076. doi: 10.1093/ptj/pzab076. PMID 33611503
- [Derived] Willaert W, Malfliet A, Coppieters I, Lenoir D, De Pauw R, Danneels L, Roussel N, Meeus M, Cagnie B, Nijs J, Kregel J. Does Pain Neuroscience Education and Cognition-Targeted Motor Control Training Improve Cervical Motor Output? Secondary Analysis of a Randomized Clinical Trial. Pain Pract. 2020 Jul;20(6):600-614. doi: 10.1111/papr.12884. Epub 2020 Apr 20. PMID 32187789
- [Derived] Lenoir D, Coppieters I, Willaert W, Kregel J, Danneels L, Cagnie B, Meeus M, Nijs J, Malfliet A. Do sociodemographic features, pain sensitivity or pain catastrophizing relate to clinic-based adherence to physiotherapy in people suffering from chronic spinal pain? Secondary analysis of a randomized clinical trial. Musculoskelet Sci Pract. 2019 Dec;44:102066. doi: 10.1016/j.msksp.2019.102066. Epub 2019 Sep 26. PMID 31605983
- [Derived] Malfliet A, Kregel J, Coppieters I, De Pauw R, Meeus M, Roussel N, Cagnie B, Danneels L, Nijs J. Effect of Pain Neuroscience Education Combined With Cognition-Targeted Motor Control Training on Chronic Spinal Pain: A Randomized Clinical Trial. JAMA Neurol. 2018 Jul 1;75(7):808-817. doi: 10.1001/jamaneurol.2018.0492. PMID 29710099
- [Derived] Malfliet A, Kregel J, Meeus M, Roussel N, Danneels L, Cagnie B, Dolphens M, Nijs J. Blended-Learning Pain Neuroscience Education for People With Chronic Spinal Pain: Randomized Controlled Multicenter Trial. Phys Ther. 2018 May 1;98(5):357-368. doi: 10.1093/ptj/pzx092. PMID 29669079
- [Derived] Dolphens M, Nijs J, Cagnie B, Meeus M, Roussel N, Kregel J, Malfliet A, Vanderstraeten G, Danneels L. Efficacy of a modern neuroscience approach versus usual care evidence-based physiotherapy on pain, disability and brain characteristics in chronic spinal pain patients: protocol of a randomized clinical trial. BMC Musculoskelet Disord. 2014 May 8;15:149. doi: 10.1186/1471-2474-15-149. PMID 24885889